CLINICAL TRIAL: NCT01537991
Title: A Phase I/II Trial of Isotoxic Accelerated Radiotherapy in the Treatment of Patients With Non-small Cell Lung Cancer
Brief Title: ISoToxic Accelerated RadioTherapy in Locally Advanced Non-small Cell Lung Cancer: The Phase I/II I-START Trial
Acronym: I-START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lisette Nixon (Other Government)
Responsible Party: Sponsor-Investigator, Lisette Nixon, Research Fellow (Senior Trial Manager in Solid Tumours), Velindre NHS Trust
Organization: Velindre NHS Trust (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/VCC/0080; ISRCTN74841904 (Other Grant/Funding Number: Cancer Research UK; CRUK/10/005)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Locally Advanced Non-small Cell Lung Cancer
Keywords: radiotherapy; non small cell lung cancer; isotoxic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1A (Experimental): Group 1A is where less than or equal to 6.5cm length of oesophagus is lying with the Planning Target Volume. Dose will be between 58 and 65Gy determined by current trial cohort in Phase I.
  Interventions: Radiation: Radiotherapy
- Group 1B (Experimental): Group 1A is where more than 6.5cm length of oesophagus is lying with the Planning Target Volume. Dose will be between 58 and 65Gy determined by current trial cohort in Phase I.
  Interventions: Radiation: Radiotherapy
- Phase II (Experimental): All patients will receive radiotherapy to a maximum dose of 65Gy in 20 fractions. The dose to the individual patient will be determined by their individual dose constraints for organs at risk.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — All patients will receive radiotherapy to the primary lung tumour and any demonstrated nodal involvement. Patients will be given radiotherapy of a dose between 58 and 65Gy in 20 fractions. Dose will be determined by the patients' group.

SUMMARY:
The I-START trial is designed to determine the highest doses of radiotherapy that can safely be used in locally advanced non-small cell lung cancer (NSCLC). Patients with NSCLC who are expected to live longer than three months and are fit to receive radical radiotherapy (radiotherapy given with curative intent) will be eligible to participate. All trial participants will receive 20 doses (called fractions) of radiotherapy. Evidence is available that suggests increasing the dose of radiotherapy given per fraction may improve both local control of the cancer and survival in some patients. However, high dose radiotherapy can damage normal tissues as well as the tumour. The dose of radiotherapy that can be used to treat lung cancer is limited by the normal tissues close to the cancer. For most of these normal tissues (lung, spinal cord and heart) the maximum safe radiotherapy dose that can be given is known. The maximum safe dose of radiotherapy for the oesophagus (gullet) is not currently known.

The trial will be split into two parts:

1. For those participants where the oesophagus will receive a high dose of radiation due to it lying close to the cancer, the first part of the trial will establish the maximum safe dose of radiotherapy to the oesophagus. The first group of participants will receive a slightly higher dose than is currently used to treat lung cancer. If these participants do not have any significant side effects, a second group of participants will receive a slightly higher dose than the first group. This process will continue incrementally until side effects from the treatment become evident, thus demonstrating the maximum dose that can safely be given. Once the maximum safe dose to the oesophagus is known this will be classed as the recommended Phase II dose and all further patients entering the trial will receive no more than this dose to the oesophagus.
2. For those participants where the cancer is a safe distance from their oesophagus, the highest dose of radiotherapy that does not exceed the known safe dose limits of the normal structures (lung, spinal cord and heart) will be used.

The findings of both parts of this study will determine whether increasing the dose of radiotherapy for NSCLC patients is a tolerable, safe and effective treatment. If the results are positive then this new treatment may be compared against the best currently available standard treatments in a future larger randomised (Phase III) trial.

DETAILED DESCRIPTION:
Main inclusion criteria:

1. Histologically or cytologically confirmed stage II - IIIb NSCLC (see appendix II)
2. Inoperable disease (as assessed by a lung cancer MDT with thoracic surgical input) or operable but the patient refuses surgery
3. Disease which can be encompassed within a radical radiotherapy treatment plan in keeping with standard practice at the participating centre
4. WHO Performance Status 0 or 1 (Appendix III)
5. Adequate respiratory function: FEV1 ≥ 1.0 litre, DLco (transfer factor) ≥ 40% of predicted and Kco (DLco/VA) > 40% predicted on baseline lung function tests
6. Blood Haemoglobin ≥ 10g/dL
7. No prior thoracic radiotherapy
8. Age ≥ 16 years
9. Considered fit to receive trial treatment
10. Estimated life expectancy of more than 3 months
11. Written informed consent obtained
12. Patient consents for electronic CT scan and planning data to be used for future research

Main exclusion criteria:

1. Medically unstable (e.g. unstable diabetes, uncontrolled hypertension, infection, hypercalcaemia or very symptomatic ischaemic heart disease)
2. Previous or current malignant disease likely to interfere with protocol treatment
3. Pancoast tumours
4. Connective tissue disorders (e.g. Scleroderma, Systemic Lupus Erythematosus)
5. Interstitial lung disease
6. Women who are pregnant or lactating
7. Women of childbearing potential who are not using adequate contraceptive precautions

   Primary outcome measure:

   Phase I:

   • Establish the maximum tolerated dose (MTD) to the oesophagus to use as the recommended Phase II dose.

   Phase II:

   • Toxicity rate (grade 3 and 4) at three months.

   Secondary outcome measures

   Phase I:

   • Chronic oesophagitis or stricture occurring/persisting two months or more after completion of radiotherapy

   Phase II:
   * Local control at three months (to include complete response, partial response and stable disease)
   * Feasibility
   * Time to Local Progression; measured in days from the day of trial entry to the date of first clinical evidence of progressive disease at the primary site
   * Time to distant metastases measured in days
   * Overall Survival; measured in days, from the day of trial entry to the day of death (from any cause)
   * Toxicity; pulmonary, oesophageal, spinal cord and cardiac grade 3 or 4 toxicity occurring up to three months after radiotherapy
   * Radiotherapy Quality Assurance. A detailed QA program will be in place to ensure adherence to the protocol. Major and minor deviations will be documented

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage II - IIIb NSCLC (see appendix II)
2. Inoperable disease (as assessed by a lung cancer MDT with thoracic surgical input) or operable but the patient refuses surgery
3. Disease which can be encompassed within a radical radiotherapy treatment plan in keeping with standard practice at the participating centre
4. WHO Performance Status 0 or 1 (Appendix III)
5. Adequate respiratory function: FEV1 ≥ 1.0 litre, DLco (transfer factor) ≥ 40% of predicted and Kco (DLco/VA) > 40% predicted on baseline lung function tests
6. Blood Haemoglobin ≥ 10g/dL
7. No prior thoracic radiotherapy
8. Age ≥ 16 years
9. Considered fit to receive trial treatment
10. Estimated life expectancy of more than 3 months
11. Written informed consent obtained
12. Patient consents for electronic CT scan and planning data to be used for future research
13. Patient is available for follow up

Exclusion Criteria:

1. Medically unstable (e.g. unstable diabetes, uncontrolled hypertension, infection, hypercalcaemia or very symptomatic ischaemic heart disease)
2. Previous or current malignant disease likely to interfere with protocol treatment
3. Pancoast tumours
4. Connective tissue disorders (e.g. Scleroderma, Systemic Lupus Erythematosus)
5. Interstitial lung disease
6. Women who are pregnant or lactating
7. Women of childbearing potential who are not using adequate contraceptive precautions

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-01-26 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Phase I: Establish the maximum tolerated dose (MTD) to the oesophagus to use as the recommended Phase II dose. | toxicity assessed up to 60 days after last Radiotherapy dose
Phase II: Toxicity rate (grade 3 and 4) at three months. | 3 months

SECONDARY OUTCOMES:
Phase I: Chronic oesophagitis or stricture occurring/persisting two months or more after completion of radiotherapy | 2 months
Pase II: Local control at three months (to include complete response, partial response and stable disease) | 3 months
Phase II: Feasibility | 2 years
Phase II: Time to Local Progression; measured in days from the day of trial entry to the date of first clinical evidence of progressive disease at the primary site | 2 years
Phase II: Time to distant metastases measured in days | 2 years
Phase II: Overall Survival; measured in days, from the day of trial entry to the day of death (from any cause) | 2 years
Phase II: Toxicity; pulmonary, oesophageal, spinal cord and cardiac grade 3 or 4 toxicity occurring up to three months after radiotherapy | 3 months
Phase II: Radiotherapy Quality Assurance. A detailed QA program will be in place to ensure adherence to the protocol. Major and minor deviations will be documented | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lester, MBBS, MRCP, FRCR, Principal Investigator — Velindre Cancer Centre; Gareth Griffiths, BSc, MSc, Cstat, Study Director — Wales Cancer Trials Unit
Locations (2):
- United Kingdom (2):
  - Velindre Cancer Centre, Cardiff, Glamorgan
  - Clatterbridge Centre for Oncology, Liverpool, Merseyside

REFERENCES:
- See also: I-START trial page — https://www.cardiff.ac.uk/centre-for-trials-research/research/studies-and-trials/view/i-start
- See also: ISRCTN database — http://www.controlled-trials.com/ISRCTN74841904
- See also: NCRI Radiotherapy Trials Quality Assurance Group — http://www.rttrialsqa.org.uk/